CLINICAL TRIAL: NCT04834102
Title: COVID-19 Induced Telogen Effluvium
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Hasan Aksoy, Specialist Dr., Istanbul Medeniyet University
Other Study IDs: 2021/0123
Record Dates: First submitted 2021-04-04; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Covid19; Telogen Effluvium; SARS-CoV Infection; Alopecia
Keywords: Telogen Effluvium; Covid-19; Alopecia
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Alopecia | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood Tests — Evaluation of blood ferritin, hemoglobine, serum iron and serum iron binding capacity

SUMMARY:
This study inquires about the development of Telogen effluvium following the SARS-CoV-2 infection

DETAILED DESCRIPTION:
Telogen effluvium (TE) is one of the most common causes of non-scarring alopecia. During the COVİD-19 pandemic, there is an increased number of Telogen effluvium patients.This study inquires about the development of Telogen effluvium following the SARS-CoV-2 infection and correlation between the severity of covid-19 and TE.

ELIGIBILITY:
Inclusion Criteria:

* Sars-CoV-2 infection in the past year

Exclusion Criteria:

* Other common causes of Telogen effluvium ( such as anemia, iron deficiency, thyroid dysfunction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults that are diagnosed with COVID-19 in the past year.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2021-04-27 (Estimated); Study Completion 2021-04-27 (Estimated)

PRIMARY OUTCOMES:
Hair shedding | 3 months
  Physical examination of hair and scalp, trichoscopy, hair pull test

CONTACTS AND LOCATIONS:
Overall Officials: Hasan AKSOY, Dr., Principal Investigator — Istanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Asghar F, Shamim N, Farooque U, Sheikh H, Aqeel R. Telogen Effluvium: A Review of the Literature. Cureus. 2020 May 27;12(5):e8320. doi: 10.7759/cureus.8320. PMID 32607303
- [Result] Mieczkowska K, Deutsch A, Borok J, Guzman AK, Fruchter R, Patel P, Wind O, McLellan BN, Mann RE, Halverstam CP. Telogen effluvium: a sequela of COVID-19. Int J Dermatol. 2021 Jan;60(1):122-124. doi: 10.1111/ijd.15313. Epub 2020 Nov 23. No abstract available. PMID 33226117
- [Result] Rizzetto G, Diotallevi F, Campanati A, Radi G, Bianchelli T, Molinelli E, Mazzanti S, Offidani A. Telogen effluvium related to post severe Sars-Cov-2 infection: Clinical aspects and our management experience. Dermatol Ther. 2021 Jan;34(1):e14547. doi: 10.1111/dth.14547. Epub 2020 Nov 23. PMID 33190397
- [Result] Cline A, Kazemi A, Moy J, Safai B, Marmon S. A surge in the incidence of telogen effluvium in minority predominant communities heavily impacted by COVID-19. J Am Acad Dermatol. 2021 Mar;84(3):773-775. doi: 10.1016/j.jaad.2020.11.032. Epub 2020 Dec 10. No abstract available. PMID 33310111